CLINICAL TRIAL: NCT05431153
Title: A PHASE 1, RANDOMIZED, OPEN-LABEL, 4-PERIOD, 5-TREATMENT, 6-SEQUENCE, CROSSOVER, SINGLE-DOSE STUDY IN HEALTHY PARTICIPANTS TO INVESTIGATE THE EFFECT OF TABLET FORMULATION AND FOOD ON THE BIOAVAILABILITY OF PF-07104091
Brief Title: A Study to Investigate the Effect of Tablet Formulation and Food on PF-07104091 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: C4161007
Record Dates: First submitted 2022-06-09; First posted 2022-06-24 (Actual); Results first posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2023-10

CONDITIONS: Healthy
Keywords: PF-07104091; Food-effect; Relative Bioavailability; Pharmacokinetics; Cyclin-Dependent Kinase 2 (CDK2) inhibitor

STUDY DESIGN:
Intervention Model Description: Randomized, open-label, 4-period, 5-treatment, 6-sequence, crossover study.
Masking Description: Open-label Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- PF-07104091 Sequence 1 (Experimental): Participants randomized to Sequence 1 will receive Treatments A, B, C, and D in Periods 1 through 4, respectively in the form of tablets by mouth.
  Interventions: Drug: Single dose of PF-07104091 as Tablet Formulation A (Treatment A); Drug: Single dose of PF-07104091 as Tablet Formulation B (Treatment B); Drug: Single dose of PF-07104091 as Tablet Formulation C (Treatment C); Drug: Single dose of PF-07104091 as Tablet Formulation D (Treatment D)
- PF-07104091 Sequence 2 (Experimental): Participants randomized to Sequence 2 will receive Treatments B, C, A, and D in Periods 1 through 4, respectively in the form of tablets by mouth.
  Interventions: Drug: Single dose of PF-07104091 as Tablet Formulation A (Treatment A); Drug: Single dose of PF-07104091 as Tablet Formulation B (Treatment B); Drug: Single dose of PF-07104091 as Tablet Formulation C (Treatment C); Drug: Single dose of PF-07104091 as Tablet Formulation D (Treatment D)
- PF-07104091 Sequence 3 (Experimental): Participants randomized to Sequence 3 will receive Treatments C, A, B, and D in Periods 1 through 4, respectively in the form of tablets by mouth.
  Interventions: Drug: Single dose of PF-07104091 as Tablet Formulation A (Treatment A); Drug: Single dose of PF-07104091 as Tablet Formulation B (Treatment B); Drug: Single dose of PF-07104091 as Tablet Formulation C (Treatment C); Drug: Single dose of PF-07104091 as Tablet Formulation D (Treatment D)
- PF-07104091 Sequence 4 (Experimental): Participants randomized to Sequence 4 will receive Treatments A, B, C, and E in Periods 1 through 4, respectively in the form of tablets by mouth.
  Interventions: Drug: Single dose of PF-07104091 as Tablet Formulation A (Treatment A); Drug: Single dose of PF-07104091 as Tablet Formulation B (Treatment B); Drug: Single dose of PF-07104091 as Tablet Formulation C (Treatment C); Drug: Single dose of PF-07104091 as Tablet Formulation C (Treatment E)
- PF-07104091 Sequence 5 (Experimental): Participants randomized to Sequence 5 will receive Treatments B, C, A, and E in Periods 1 through 4, respectively in the form of tablets by mouth.
  Interventions: Drug: Single dose of PF-07104091 as Tablet Formulation A (Treatment A); Drug: Single dose of PF-07104091 as Tablet Formulation B (Treatment B); Drug: Single dose of PF-07104091 as Tablet Formulation C (Treatment C); Drug: Single dose of PF-07104091 as Tablet Formulation C (Treatment E)
- PF-07104091 Sequence 6 (Experimental): Participants randomized to Sequence 6 will receive Treatments C, A, B, and E in Periods 1 through 4, respectively in the form of tablets by mouth.
  Interventions: Drug: Single dose of PF-07104091 as Tablet Formulation A (Treatment A); Drug: Single dose of PF-07104091 as Tablet Formulation B (Treatment B); Drug: Single dose of PF-07104091 as Tablet Formulation C (Treatment C); Drug: Single dose of PF-07104091 as Tablet Formulation C (Treatment E)

INTERVENTIONS:
Drug: Single dose of PF-07104091 as Tablet Formulation A (Treatment A) — A single dose of PF-07104091 as Tablet Formulation A administered under fasting conditions.
  Other Names: Tablet Formulation A, Fasted
Drug: Single dose of PF-07104091 as Tablet Formulation B (Treatment B) — A single dose of PF-07104091 as Tablet Formulation B administered under fasting conditions.
  Other Names: Tablet Formulation B, Fasted
Drug: Single dose of PF-07104091 as Tablet Formulation C (Treatment C) — A single dose of PF-07104091 as Tablet Formulation C administered under fasting conditions.
  Other Names: Tablet Formulation C, Fasted
Drug: Single dose of PF-07104091 as Tablet Formulation D (Treatment D) — A single dose of PF-07104091 as Tablet Formulation D administered under fasting conditions.
  Other Names: Tablet Formulation D, Fasted
  Arms: PF-07104091 Sequence 1; PF-07104091 Sequence 2; PF-07104091 Sequence 3
Drug: Single dose of PF-07104091 as Tablet Formulation C (Treatment E) — A single dose of PF-07104091 as Tablet Formulation C administered under fed conditions.
  Other Names: Tablet Formulation C, Fed
  Arms: PF-07104091 Sequence 4; PF-07104091 Sequence 5; PF-07104091 Sequence 6

SUMMARY:
This is a single dose crossover pharmacokinetic (pharmacokinetics helps in understanding how the drug is changed and eliminated from the body after a participant takes it) study in healthy participants. The study consists of 5 treatments, and each participant will be randomized to receive 4 of the treatments in separate periods in a specific sequence. Each treatment consists of a single dose of PF-07104091 and the treatments differ by tablet formulation and/or whether the dose is to be given under fasted or fed conditions. Plasma pharmacokinetics of PF-07104091 will be assessed following each dose to determine the effect of tablet formulation and fed condition on the relative bioavailability of PF-07104091.

ELIGIBILITY:
Inclusion Criteria:

* Male participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, vital signs, and standard 12 lead ECGs.
* Body-Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight of >50 kg (110 lb).
* Written evidence of a personally signed and dated informed consent document (ICD) indicating that the participant has been informed of all pertinent aspects of the study.
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
* History of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HBsAg), Hepatitis B core antibody (HBcAB) or hepatitis C antibody (HCVAb). Hepatitis B vaccination is allowed.
* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions or situations related to COVID-19 pandemic (eg, contact with positive case, residence, or travel to an area with high incidence) that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention.
* A positive urine drug test.
* History of sensitivity to heparin or heparin induced thrombocytopenia.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2022-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4161007

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 30 participants were randomly assigned and received the study treatment.
Groups:
- Treatment Sequence ABCD: Participants received a single 300 milligrams (mg) dose (2*125 mg and 2*25 mg) of PF-07104091 tablet Formulation A under fasting conditions (Treatment A) on Day 1 of period 1 followed by 300 mg (2*125 mg and 2*25 mg) tablet Formulation B under fasting condition (Treatment B) on Day 1 of period 2 followed by 300 mg (4*75 mg) tablet Formulation C under fasting condition (Treatment C) on Day 1 of period 3 followed by 300 mg (4*75 mg) tablet Formulation D under fasting condition (Treatment D) on Day 1 of period 4. There was a washout period of 5 days between each treatment period.
- Treatment Sequence BCAD: Participants received a single 300 mg (2*125 mg and 2*25 mg) PF-07104091 tablet Formulation B under fasting condition (Treatment B) on Day 1 of period 1 followed by 300 mg (4*75 mg) tablet Formulation C under fasted condition (Treatment C) on Day 1 of treatment period 2 followed by 300 mg (2*125 mg and 2*25 mg) tablet Formulation A under fasting condition (Treatment A) on Day 1 of period 3 followed by 300 mg (4*75 mg) tablet Formulation D under fasted condition (Treatment D) on Day 1 of period 4. There was a washout period of 5 days between each treatment period.
- Treatment Sequence CABD: Participants received a single 300 mg (4*75 mg) PF-07104091 tablet Formulation C under fasting condition (Treatment C) on Day 1 of period 1 followed by 300 mg (2*125 mg and 2*25 mg) tablet Formulation A under fasting condition (Treatment A) on Day 1 of period 2 followed by 300 mg (2*125 mg and 2*25 mg) tablet Formulation B under fasting condition (Treatment B) on Day 1 of period 3 followed by 300 mg (4*75 mg) tablet Formulation D under fasting condition (Treatment D) on Day 1 of period 4. There was a washout period of 5 days between each treatment period.
- Treatment Sequence ABCE: Participants received a single 300 mg (2*125 mg and 2*25 mg) PF-07104091 tablet Formulation A under fasting condition (Treatment A) on Day 1 of period 1 followed by 300 mg (2*125 mg and 2*25 mg) tablet Formulation B under fasting condition (Treatment B) on Day 1 of period 2 followed by 300 mg (4*75 mg) tablet Formulation C under fasting condition (Treatment C) on Day 1 of period 3 followed by 300 mg (4*75 mg) tablet Formulation C under fed condition (Treatment E) on Day 1 of period 4. There was a washout period of 5 days between each treatment period.
- Treatment Sequence BCAE: Participants received a single 300 mg (2*125 mg and 2*25 mg) PF-07104091 tablet Formulation B under fasting condition (Treatment B) on Day 1 of period 1 followed by 300 mg (4*75 mg) tablet Formulation C under fasting condition (Treatment C) on Day 1 of period 2 followed by 300 mg (2*125 mg and 2*25 mg) tablet Formulation A under fasting condition (Treatment A) on Day 1 of period 3 followed by 300 mg (4*75 mg) tablet Formulation C under fed condition (Treatment E) on Day 1 of period 4. There was a washout period of 5 days between each treatment period.
- Treatment Sequence CABE: Participants received a single 300 mg (4*75 mg) PF-07104091 tablet Formulation C under fasting condition (Treatment C) on Day 1 of period 1 followed by 300 mg (2*125 mg and 2*25 mg) tablet Formulation A under fasting condition (Treatment A) on Day 1 of period 2 followed by 300 mg (2*125 mg and 2*25 mg) tablet Formulation B under fasting condition (Treatment B) on Day 1 of period 3 followed by 300 mg (4*75 mg) tablet Formulation C under fed condition (Treatment E) on Day 1 of period 4. There was a washout period of 5 days between each treatment period.
Period: Treatment Period 1 (Day 1)
Arm/Group | Treatment Sequence ABCD | Treatment Sequence BCAD | Treatment Sequence CABD | Treatment Sequence ABCE | Treatment Sequence BCAE | Treatment Sequence CABE
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 4 | 5
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0
Period: Washout Period 1 (5 Days)
Arm/Group | Treatment Sequence ABCD | Treatment Sequence BCAD | Treatment Sequence CABD | Treatment Sequence ABCE | Treatment Sequence BCAE | Treatment Sequence CABE
Started | 5 | 5 | 5 | 5 | 4 | 5
Completed | 5 | 5 | 5 | 5 | 4 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2 (Day 1)
Arm/Group | Treatment Sequence ABCD | Treatment Sequence BCAD | Treatment Sequence CABD | Treatment Sequence ABCE | Treatment Sequence BCAE | Treatment Sequence CABE
Started | 5 | 5 | 5 | 5 | 4 | 5
Completed | 5 | 5 | 5 | 5 | 4 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 2 (5 Days)
Arm/Group | Treatment Sequence ABCD | Treatment Sequence BCAD | Treatment Sequence CABD | Treatment Sequence ABCE | Treatment Sequence BCAE | Treatment Sequence CABE
Started | 5 | 5 | 5 | 5 | 4 | 5
Completed | 5 | 5 | 5 | 5 | 4 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 3 (Day 1)
Arm/Group | Treatment Sequence ABCD | Treatment Sequence BCAD | Treatment Sequence CABD | Treatment Sequence ABCE | Treatment Sequence BCAE | Treatment Sequence CABE
Started | 5 | 5 | 5 | 5 | 4 | 5
Completed | 5 | 5 | 5 | 5 | 4 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 3 (5 Days)
Arm/Group | Treatment Sequence ABCD | Treatment Sequence BCAD | Treatment Sequence CABD | Treatment Sequence ABCE | Treatment Sequence BCAE | Treatment Sequence CABE
Started | 5 | 5 | 5 | 5 | 4 | 5
Completed | 5 | 5 | 5 | 5 | 4 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 4 (Day 1)
Arm/Group | Treatment Sequence ABCD | Treatment Sequence BCAD | Treatment Sequence CABD | Treatment Sequence ABCE | Treatment Sequence BCAE | Treatment Sequence CABE
Started | 5 | 5 | 5 | 5 | 4 | 5
Completed | 5 | 5 | 5 | 5 | 4 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants were analyzed.
Groups:
- Treatment Sequence ABCD+BCAD+CABD: All participants who received Treatment A: PF-07104091 300 mg (2*125 mg and 2*25 mg) tablet Formulation A, under fasting condition, treatment B: 300 mg (2*125 mg and 2*25 mg) tablet Formulation B under fasting condition, treatment C: 300 mg (4*75 mg) tablet Formulation C under fasting condition, treatment D: 300 mg (4*75 mg) tablet Formulation D under fasting condition, in either Period 1, 2, 3, and 4 based on the treatment sequence were included.
- Treatment Sequence ABCE+BCAE+CABE: All participants who received Treatment A: PF-07104091 300 mg (2*125 mg and 2*25 mg) tablet Formulation A, under fasting condition, treatment B: 300 mg (2*125 mg and 2*25 mg) tablet Formulation B, under fasting condition, treatment C: 300 mg (4*75 mg) tablet Formulation C under fasting condition, treatment E: 300 mg (4*75 mg) tablet Formulation C under fed condition in either Period 1, 2, 3, and 4 based on the treatment sequence were included.
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence ABCD+BCAD+CABD | Treatment Sequence ABCE+BCAE+CABE | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.9 (13.04) | 40.3 (13.06) | 41.1 (12.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 15 | 15 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 13 | 10 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 8 | 14
  White | 6 | 7 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma-Concentration Time Curve From Time Zero (0) Extrapolated to Infinity (AUCinf) of PF-07104091 for Treatment A, B, and C
Description: AUCinf was calculated as AUClast + (Clast/kel) where Clast was the predicted plasma concentration at the last quantifiable time point from the log-linear regression analysis and kel was the terminal phase rate constant calculated by a linear regression of the log linear concentration-time curve.
Time Frame: Predose, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, and 48 hours post-dose
Population: Pharmacokinetic (PK) Parameter set included all participants randomized and treated who had at least 1 of the PF-07104091 PK parameters of primary interest in at least 1 treatment period. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms*hour per milliliter
Groups:
- Treatment A: PF-07104091 Tablet Formulation A (Fasted): Participants received a single 300 mg dose (2*125 mg and 2*25 mg) of PF-07104091 tablet Formulation A, under fasting conditions.
- Treatment B: PF-07104091 Tablet Formulation B (Fasted): Participants received a single 300 mg dose (2*125 mg and 2*25 mg) of PF-07104091 tablet Formulation B, under fasting conditions.
- Treatment C: PF-07104091 Tablet Formulation C (Fasted): Participants received a single 300 mg dose (4*75 mg) of PF-07104091 tablet Formulation C, under fasting conditions.
Arm/Group | Treatment A: PF-07104091 Tablet Formulation A (Fasted) | Treatment B: PF-07104091 Tablet Formulation B (Fasted) | Treatment C: PF-07104091 Tablet Formulation C (Fasted)
Number analyzed (Participants) | 21 | 18 | 19
Nanograms*hour per milliliter | 10920 (34) | 10720 (28) | 11200 (32)
Statistical Analysis 1: Comparison: Treatment A: PF-07104091 Tablet Formulation A (Fasted) vs Treatment B: PF-07104091 Tablet Formulation B (Fasted); Test type: Other; Ratio of adjusted geometric means = 98.83, 90% CI 2-sided [94.00 to 103.91] — Values were back-transformed from the log scale. The model was a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect
Statistical Analysis 2: Comparison: Treatment A: PF-07104091 Tablet Formulation A (Fasted) vs Treatment C: PF-07104091 Tablet Formulation C (Fasted); Test type: Other; Ratio of adjusted geometric means = 98.02, 90% CI 2-sided [93.88 to 102.35] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Treatment B: PF-07104091 Tablet Formulation B (Fasted) vs Treatment C: PF-07104091 Tablet Formulation C (Fasted); Test type: Other; Ratio of adjusted geometric means = 98.51, 90% CI 2-sided [91.79 to 105.73] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-07104091 for Treatment A, B and C
Description: Cmax was maximum observed concentration. Cmax was observed directly from data.
Time Frame: Predose, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, and 48 hours post-dose
Population: PK Parameter set included all participants randomized and treated who had at least 1 of the PF-07104091 PK parameters of primary interest in at least 1 treatment period. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Treatment A: PF-07104091 Tablet Formulation A (Fasted) | Treatment B: PF-07104091 Tablet Formulation B (Fasted) | Treatment C: PF-07104091 Tablet Formulation C (Fasted)
Number analyzed (Participants) | 27 | 28 | 27
Nanograms per milliliter | 1531 (31) | 1490 (28) | 1415 (34)
Statistical Analysis 1: Comparison: Treatment A: PF-07104091 Tablet Formulation A (Fasted) vs Treatment B: PF-07104091 Tablet Formulation B (Fasted); Test type: Other; Ratio of adjusted geometric means = 96.35, 90% CI 2-sided [87.48 to 106.12] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Treatment A: PF-07104091 Tablet Formulation A (Fasted) vs Treatment C: PF-07104091 Tablet Formulation C (Fasted); Test type: Other; Ratio of adjusted geometric means = 93.47, 90% CI 2-sided [85.65 to 102.00] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Treatment B: PF-07104091 Tablet Formulation B (Fasted) vs Treatment C: PF-07104091 Tablet Formulation C (Fasted); Test type: Other; Ratio of adjusted geometric means = 98.01, 90% CI 2-sided [89.86 to 106.90] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: AUCinf of PF-07104091 for Treatment C, D and E
Description: as for outcome 1
Time Frame: Predose, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, and 48 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms*hour per milliliter
Groups:
- Treatment D: PF-07104091 Tablet Formulation D (Fasted): Participants received a single 300 mg dose (4*75 mg) of PF-07104091 tablet Formulation D, under fasting conditions.
- Treatment E: PF-07104091 Tablet Formulation C (Fed): Participants received a single 300 mg dose (4*75 mg) of PF-07104091 tablet Formulation C, given with a high-fat/high-calorie meal.
Arm/Group | Treatment C: PF-07104091 Tablet Formulation C (Fasted) | Treatment D: PF-07104091 Tablet Formulation D (Fasted) | Treatment E: PF-07104091 Tablet Formulation C (Fed)
Number analyzed (Participants) | 19 | 10 | 11
Nanograms*hour per milliliter | 11200 (32) | 12850 (32) | 10500 (24)
Statistical Analysis 1: Comparison: Treatment C: PF-07104091 Tablet Formulation C (Fasted) vs Treatment D: PF-07104091 Tablet Formulation D (Fasted); Test type: Other; Ratio of adjusted geometric means = 111.52, 90% CI 2-sided [99.55 to 124.93] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Treatment C: PF-07104091 Tablet Formulation C (Fasted) vs Treatment E: PF-07104091 Tablet Formulation C (Fed); Test type: Other; Ratio of adjusted geometric means = 98.38, 90% CI 2-sided [90.68 to 106.73] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Cmax of PF-07104091 for Treatment C, D and E
Description: Cmax was maximum observed concentration. Cmax was observed directly from data.
Time Frame: Predose, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, and 48 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Groups:
- Treatment C: PF-07104091 Tablet Formulation (Fasted): Participants received a single 300 mg dose (4*75 mg) of PF-07104091 tablet Formulation C, under fasting conditions.
Arm/Group | Treatment C: PF-07104091 Tablet Formulation (Fasted) | Treatment D: PF-07104091 Tablet Formulation D (Fasted) | Treatment E: PF-07104091 Tablet Formulation C (Fed)
Number analyzed (Participants) | 27 | 13 | 14
Nanograms per milliliter | 1415 (34) | 1498 (36) | 1193 (36)
Statistical Analysis 1: Comparison: Treatment C: PF-07104091 Tablet Formulation (Fasted) vs Treatment D: PF-07104091 Tablet Formulation D (Fasted); Test type: Other; Ratio of adjusted geometric means = 111.52, 90% CI 2-sided [96.46 to 128.93] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Treatment C: PF-07104091 Tablet Formulation (Fasted) vs Treatment E: PF-07104091 Tablet Formulation C (Fed); Test type: Other; Ratio of adjusted geometric means = 81.39, 90% CI 2-sided [75.06 to 88.26] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. A serious adverse event (SAE) was defined as any untoward medical occurrence that, at any dose, met one or more of the following criteria: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a suspected transmission via a Pfizer product of an infectious agent, pathogenic or non-pathogenic, other important medical events. TEAEs were defined as events that occurred after start of treatment.
Time Frame: From start of study treatment until 35 days after last dose of study treatment (Up to Day 54)
Population: Safety analysis set included all participants randomly assigned to study intervention and who received at least 1 dose of study intervention. Participants were analyzed according to the study intervention they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: PF-07104091 Tablet Formulation A (Fasted) | Treatment B: PF-07104091 Tablet Formulation B (Fasted) | Treatment C: PF-07104091 Tablet Formulation C (Fasted) | Treatment D: PF-07104091 Tablet Formulation D (Fasted) | Treatment E: PF-07104091 Tablet Formulation C (Fed)
Number analyzed (Participants) | 29 | 30 | 29 | 15 | 14
Participants
  TEAEs | 21 | 19 | 17 | 7 | 2
  Serious TEAEs | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Clinical hematology parameters included: hemoglobin, hematocrit, red blood cell count, platelet count, white blood cell count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes; chemistry parameters included: blood urea nitrogen and creatinine, cystatin C and estimated glomerular filtration rate, glucose (fasting), calcium, sodium, potassium, chloride, total bicarbonate, aspartate aminotransferase, alanine aminotransferase, total bilirubin, alkaline phosphatase, uric acid, albumin, total protein, urinalysis parameters included: local dipstick: potential of hydrogen (pH), glucose, protein, blood, ketones, nitrites, leukocyte esterase. Number of participants with abnormal findings are presented in this outcome measure.
Time Frame: From start of study treatment until 35 days after last dose of study treatment (Up to Day 54)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: PF-07104091 Tablet Formulation A (Fasted) | Treatment B: PF-07104091 Tablet Formulation B (Fasted) | Treatment C: PF-07104091 Tablet Formulation C (Fasted) | Treatment D: PF-07104091 Tablet Formulation D (Fasted) | Treatment E: PF-07104091 Tablet Formulation C (Fed)
Number analyzed (Participants) | 29 | 30 | 29 | 15 | 14
Participants | 0 | 0 | 1 | 3 | 1

7. Secondary Outcome: Number of Participants With Clinically Meaningful Findings in Electrocardiogram (ECG) Assessments
Description: A 12-lead ECG was performed. Clinically meaningful findings in ECG assessments were based on the investigator's judgment.
Time Frame: From start of study treatment until 35 days after last dose of study treatment (Up to Day 54)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: PF-07104091 Tablet Formulation A (Fasted) | Treatment B: PF-07104091 Tablet Formulation B (Fasted) | Treatment C: PF-07104091 Tablet Formulation C (Fasted) | Treatment D: PF-07104091 Tablet Formulation D (Fasted) | Treatment E: PF-07104091 Tablet Formulation C (Fed)
Number analyzed (Participants) | 29 | 30 | 29 | 15 | 14
Participants | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Clinically Meaningful Findings in Vital Signs
Description: Vital signs were measured with the participant's arm supported at the level of the heart after approximately 5 minutes of rest. Vital signs parameters included: diastolic and systolic blood pressure, respiratory rate, pulse rate, and temperature. Number of participants with clinically meaningful findings in any vital sign parameter were reported. Clinically meaningful findings were based on the investigator's judgment.
Time Frame: From start of study treatment until 35 days after last dose of study treatment (Up to Day 54)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: PF-07104091 Tablet Formulation A (Fasted) | Treatment B: PF-07104091 Tablet Formulation B (Fasted) | Treatment C: PF-07104091 Tablet Formulation C (Fasted) | Treatment D: PF-07104091 Tablet Formulation D (Fasted) | Treatment E: PF-07104091 Tablet Formulation C (Fed)
Number analyzed (Participants) | 29 | 30 | 29 | 15 | 14
Participants | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Clinically Meaningful Findings in Physical Examination Assessments
Description: A complete physical examination included at a minimum, head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, and gastrointestinal, musculoskeletal, and neurological systems. A brief physical examination included at a minimum, assessments of general appearance, the respiratory and cardiovascular systems, and participant-reported symptoms. Clinically significant findings were defined according to investigator's assessment.
Time Frame: From start of study treatment until 35 days after last dose of study treatment (Up to Day 54)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: PF-07104091 Tablet Formulation A (Fasted) | Treatment B: PF-07104091 Tablet Formulation B (Fasted) | Treatment C: PF-07104091 Tablet Formulation C (Fasted) | Treatment D: PF-07104091 Tablet Formulation D (Fasted) | Treatment E: PF-07104091 Tablet Formulation C (Fed)
Number analyzed (Participants) | 29 | 30 | 29 | 15 | 14
Participants | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of study treatment until 35 days after last dose of study treatment (Up to Day 54)
Description: Analysis was performed on safety analysis set.
Arm/Group | Treatment A: PF-07104091 Tablet Formulation A (Fasted) | Treatment B: PF-07104091 Tablet Formulation B (Fasted) | Treatment C: PF-07104091 Tablet Formulation C (Fasted) | Treatment D: PF-07104091 Tablet Formulation D (Fasted) | Treatment E: PF-07104091 Tablet Formulation C (Fed)
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/30 | 0/29 | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30 | 0/29 | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 21/29 | 18/30 | 17/29 | 7/15 | 2/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Treatment A: PF-07104091 Tablet Formulation A (Fasted) (N=29) | Treatment B: PF-07104091 Tablet Formulation B (Fasted) (N=30) | Treatment C: PF-07104091 Tablet Formulation C (Fasted) (N=29) | Treatment D: PF-07104091 Tablet Formulation D (Fasted) (N=15) | Treatment E: PF-07104091 Tablet Formulation C (Fed) (N=14)
Breath odour (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 4 | 5 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0
Eructation (Gastrointestinal disorders) | 2 | 0 | 0/20 | 0 | 0
Nausea (Gastrointestinal disorders) | 18/20 | 14 | 13 | 4 | 1
Vomiting (Gastrointestinal disorders) | 6 | 7 | 3 | 3 | 0
Chills (General disorders) | 2 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 3 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0/20 | 0 | 0 | 1 | 0
Appetite disorder (Metabolism and nutrition disorders) | 0/20 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 3 | 1 | 3 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 3 | 5 | 3 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-04-21): https://cdn.clinicaltrials.gov/large-docs/53/NCT05431153/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-09): https://cdn.clinicaltrials.gov/large-docs/53/NCT05431153/SAP_001.pdf